CLINICAL TRIAL: NCT03923166
Title: Pyrotinib Combined With Capecitabine Metronomic Therapy in HER2-postitive Advanced Breast Cancer: Single Arm, Single Center, Phase II Clinical Trial.
Brief Title: Pyrotinib Combined With Capecitabine Metronomic Therapy in HER2-postitive Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Li Qiao, Clinical Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LQ006
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pyrotinib+ capecitabine (Experimental)
  Interventions: Drug: Pyrotinib; Drug: capecitabine

INTERVENTIONS:
Drug: Pyrotinib — 400mg qd
Drug: capecitabine — capecitabine 500mg tid

SUMMARY:
Overexpression of the HER2 gene accounts for 20% to 30% of breast cancer. Although trastuzumab combined with chemotherapy has become the basic treatment for patients with HER2-positive advanced breast cancer, For patients who have progressed or relapsed after trastuzumab treatment, There are still many issues to explore on the choice of program of retargeted therapy. In HER2-positive advanced breast cancer, the results of Phase I and Phase I/II trials of pyrotinib or pyrotinib combined with capecitabine show that the anti-tumor effect is rapid, efficient and sustainable, and the patient is safe and well tolerated. Capecitabine is an oral cytotoxic drug that has high selectivity and specificity against tumors. Many patients need to adjust the dose due to adverse reactions, especially for patients after multi-line treatment. Previous studies have shown that sustained low-dose capecitabine reduces the adverse effects of the drug while ensuring efficacy. Based on the above, this study is to conduct a single-center, one-arm phase II clinical trial to explore the efficacy and safety of pyrotinib and capecitabine in the treatment of HER2-positive advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age：18~75 years;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
3. A life expectancy of more than 12 weeks;
4. patients have at least one measurable lesion exists according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria and progresses after the last anti-tumor treatment or during treatment;
5. Pathologically confirmed HER2-expressing patients with locally advanced or metastatic breast cancer: HER2 IHC 3+, or HER2 IHC 2+ and FISH detection gene amplification
6. Progression after treatment with trastuzumab (receiving at least 6 weeks of trastuzumab treatment);
7. Have not received capecitabine for the past, or Previously received capecitabine and PFS for more than 6 months;
8. echocardiography indicates that LVEF ≥ 50%;
9. The laboratory tests confirmed that the bone marrow function and liver and kidney function of the patient met the following requirements before the first dose:

   1. ANC≥1.5×10^9/L；
   2. PLT≥100×10^9/L;
   3. Hb≥100 g/L
   4. serum creatinine(Scr) less than 1.5 times the upper limit of normal value or the creatinine clearance rate calculated greater than 60 mL/min;
   5. total bilirubin less than 1.5 times the upper limit of normal value
   6. aspartate aminotransferase (AST), or alanine aminotransferase (ALT) less than 2.5 times the upper limit of normal value, less than 5 times the upper limit of normal value in patients with liver metastases;
   7. urine routine test with urinary protein more than ++, or 24 hour urinary protein more than 1.0 g;
10. Females of childbearing potential must be a pregnancy test in 7 days before participating ( including serum or urine), and the results were negative, and they are willing to take effective contraceptive methods during the trial;
11. The patient volunteered to join the study and signed an informed consent form.

Exclusion Criteria:

1. Patients who have been treated with capecitabine for a period of 6 months and whose disease progresses;
2. Previously treated with pyrotinib or neratinib;
3. Patients with high blood pressure who are not well controlled by antihypertensive medication (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg); have uncontrolled or severe cardiovascular disease, such as within 6 months before screening Refractory angina pectoris, congestive heart failure occurred; myocardial infarction occurred within 12 months before screening; any clinically significant ventricular arrhythmia history, QT interval prolongation; history of cerebrovascular accident, symptomatic and need Medically treated coronary heart disease;
4. having significant clinical dysfunction of the digestive tract may affect the intake, transport or absorption of oral medications (eg, inability to swallow, chronic diarrhea, intestinal obstruction, etc.)
5. Refractory, 2 degrees and above persistent diarrhea;
6. exiting unstable brain metastasis and / or meningeal metastasis;
7. Have undergone major surgery or severe traumatic injury, fracture, or healed wound within 4 weeks;
8. Allergic to pyrotinib, capecitabine and/or its excipients has been confirmed;
9. Female patients during pregnancy or lactation, female patients with fertility and positive pregnancy test, or women of childbearing age who are unwilling to take effective contraceptive measures during the whole trial period;
10. The patient has a severe concomitant disease, or any other condition that the investigator believes is not suitable for the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-04-19 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | 4 months
  Refers to the proportion of patients whose tumors have shrunk to a certain proportion and maintained for a certain period of time, including cases of CR and PR, RECIST 1.1 were used to assess objective tumor remission

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | 4 months
  the date from the first dose to the first occurrence of disease progression or death from any cause, whichever occurs first

OTHER OUTCOMES:
disease control rate(DCR) | 4 months
  Percentage of confirmed complete remission (CR), partial remission (PR), and disease stable (SD) cases in patients with evaluable efficacy
Incidence of adverse events | 1 Month
  safety

CONTACTS AND LOCATIONS:
Overall Officials: Qiao Li, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Binghe Xu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided